CLINICAL TRIAL: NCT04774926
Title: One Year, Single Arm, Open Label, Multicenter, Phase IV Study Using Multimodal Imaging to Guide Disease Activity Assessment Through Innovative Early Predictive Anatomical Biomarkers of Fluid Resolution in wAMD Patients Treated With Brolucizumab- IMAGINE Study
Brief Title: Study of Innovative Multimodal Imaging Biomarkers to Predict Anatomical Outcome in Naive Patients With wAMD Treated With Brolucizumab.
Acronym: IMAGINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258AIT04; 2020-002452-20 (EudraCT Number)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular age-related macular degeneration; anti-VEGF; brolucizumab; choroidal neovascularization; multimodal imaging biomarkers; fluid resolution; Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; AMD
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: The study is a one-year, open-label, single arm, multicenter, phase IV study in patients with wAMD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brolucizumab 6 mg (Experimental): Participants received 3 monthly ocular injections followed by a q12w or q8w maintenance phase based on patient's disease activity (DA).
  Interventions: Drug: Brolucizumab

INTERVENTIONS:
Drug: Brolucizumab — 120 mg/ml solution for intravitreal injection
  Other Names: RTH258, Beovu

SUMMARY:
The purpose of this study was to identify innovative early imaging parameters as predictors of the long-term clinical response to brolucizumab in terms of fluid resolution in patients with wet Age-related Macular Degeneration (wAMD) to evaluate their potential in supporting the choice of treatment regimen (q12w or q8w).

DETAILED DESCRIPTION:
The study was a one-year, open-label, single arm, multicenter, phase IV study in patients with wAMD. The study planned to enroll approximately 263 (male and female) patients aged 50 years or older with untreated active subfoveal choroidal neovascularization (CNV) secondary to wAMD in the study eye from approximately 30 centers in Italy. The duration of the study treatment for enrolled patients was a maximum of 48 weeks, consisting of 8 weeks of three monthly loading doses and 40 weeks of maintenance regimen period (q8w or q12w) according to disease activity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained prior to participation in the study
* Active choroidal neo-vascularization (CNV) secondary to AMD that affects the central subfield, including retinal angiomatous proliferation (RAP) with a CNV component, confirmed by presence of active leakage from CNV seen by fluorescein angiography (or other imaging modalities) and sequelae of CNV, e.g. pigment epithelial detachment (PED), subretinal or sub-retinal pigment epithelium (sub-RPE) hemorrhage, blocked fluorescence, macular edema in the study eye at Screening;
* Presence of intraretinal fluid (IRF) or subretinal fluid (SRF) affecting the central subfield (study eye), as seen by SD-OCT in the study eye at Screening;
* Best-corrected visual acuity (BCVA) score greater than or equal to 23 letters measured at 4-meters starting distance using Early Treatment Diabetic Retinopathy Study (EDTRS) visual acuity charts at both Screening and Baseline visits in the study eye.

Exclusion Criteria:

* Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis) in study eye at Screening or Baseline;
* Not interpretable OCTA and SD-OCT images according to Investigator's clinical judgment at Screening in the study eye;
* Concomitant conditions or ocular disorders in the study eye, at Screening or Baseline which, in the opinion of the Investigator, could prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the course of the study;
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication or according to Investigator's judgment at Screening or Baseline;
* Previous treatment with any anti-vascular endothelial growth factor (anti-Vascular endothelial growth factor (VEGF)) drugs or investigational drugs (other than vitamin supplements) in the study eye at any time prior to Screening;
* Systemic anti-VEGF therapy at any time;
* Stroke or myocardial infarction in the 6-month period prior to Baseline.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Italy (14):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Lupidi M, Bandello F, Vujosevic S, Parravano M, Bacherini D, Minnella AM, Giansanti F, Ascardi C, Staurenghi G. Multimodal Imaging to Assess Disease Activity and Predict Fluid Resolution in Patients with wAMD Treated with Brolucizumab: The IMAGINE Study. Ophthalmol Ther. 2025 Oct;14(10):2497-2510. doi: 10.1007/s40123-025-01229-5. Epub 2025 Aug 20. PMID 40833455
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2316

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If both eyes were eligible as per the inclusion and exclusion criteria, only one eye was treated during the study, with the eye with the worse visual acuity (BCVA) at Baseline selected as the study eye. If both eyes had the same BCVA, the right eye was chosen as the study eye.
Period: Overall Study
Arm/Group | Brolucizumab 6 mg
Started | 122
Completed | 91
Not Completed | 31
Not completed — Adverse Event | 15
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 3
Not completed — The original PI resigned and a new one could not be appointed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.1 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 122
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Classified as q12w Fluid-free or Not q12w Fluid-free
Description: Early predictive factors of fluid-free response is defined as the absence of retinal fluid at Week 48 in patients with a stable q12w treatment regimen up to Week 48 after the loading phase, As assessed by Spectral Domain Optical Coherence Tomography (SD-OCT).
  q12w fluid-free: pts completing the treatment and the study maintaining a stable q12w regimen assigned at Wk 16 up to Wk 48 and without the presence of IRF and SRF at Wk 48.
  not q12w fluid-free:
  * Pt who completed treatment and the study with the presence of IRF or SRF at Wk 48
  * Pt who followed the q8w regimen of treatment at any time during the study (considering also who started with q12w regimen but then due to disease activity shifted to q8w regimen)
  * Pt who discontinued treatment at any time after b/l since treatment disc. was considered as intercurrent event and a 'failure'.
  * Pt who dropped out at any time after b/l since study disc. was considered as intercurrent event and a 'failure'.
Time Frame: Up to Week 48
Population: Full Analysis Set - includes all patients who received at least one dose of the study drug and with a valid measurement without a protocol deviation with impact. (Excludes patients with protocol deviations.)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 120
Participants
  q12w fluid free - NO | 93
  q12w fluid free - YES | 27

2. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Type of Predominant Basal Choroidal Neovascularization (CNV) Lesion Type, as Assessed by SD-OCT at Baseline - Patients Classified as Not q12w Fluid-free
Description: As assessed by Spectral Domain Optical Coherence Tomography (SD-OCT).
  Percentages were computed on Safety Population within 'No' and 'Yes' groups according to q12w fluid free.
  Type 1 neovascularization arises when CNV proliferation occurs below the Retinal Pigment Epithelium (RPE) and corresponds to occult CNV with a poorly defined pattern of leakage on fluorescein angiography (FA). Type 2 neovascularization refers to CNV proliferation above the RPE in the subretinal space and corresponds to classic CNV with intense fluorescein leakage. Type 3 neovascularization (or retinal angiomatous proliferation [RAP]) occurs when retinal circulation is involved, with an anastomosis between the choroidal and retinal circulations.
  Types 1-3 classification is a classification according to the type of anatomical lesion and is determined by multimodal imaging characteristics. Please note that by design, this is not a grading nor scores on a scale.
  PCV = Polypoidal Choroidal Vasculopathy
Time Frame: Baseline
Population: Full Analysis Set - includes all patients who received at least one dose of the study drug and with a valid measurement without a protocol deviation with impact and who were classified as not q12w fluid-free (N=93). (Excludes patients with protocol deviations.)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  TYPE I + PCV; q12w fluid free - No | 61
  TYPE II; q12w fluid free - No | 21
  TYPE III; q12w fluid free - No | 5
  Missing; q12w fluid free - No | 6

3. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Type of Predominant Basal Choroidal Neovascularization (CNV) Lesion Type, as Assessed by SD-OCT at Baseline - Patients Classified as q12w Fluid-free
Description: as for outcome 2
Time Frame: Baseline
Population: Full Analysis Set - includes all patients who received at least one dose of the study drug and with a valid measurement without a protocol deviation with impact and who were classified as q12w fluid-free (N=27). (Excludes patients with protocol deviations.)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  TYPE I + PCV; q12w fluid free - Yes | 19
  TYPE II; q12w fluid free - Yes | 4
  TYPE III; q12w fluid free - Yes | 3
  Missing; q12w fluid free- Yes | 1

4. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Sub-retinal Pigment Epithelium (Sub-RPE) Fluid - Patients Classified as Not q12w Fluid-free
Description: As assessed by Spectral Domain Optical Coherence Tomography (SD-OCT).
  Percentages were computed on Safety Population within 'No' and 'Yes' groups according to q12w fluid free.
  Of note, the category 'Stable absent' is considered also for cases with baseline and last measurement collected equal to 'No' even if there are at least one 'Yes' in one of the other collected measurements. Similarly, the category 'Stable present' is considered also for cases with baseline and last measurement collected equal to 'Yes' even if there are at least one 'No' in one of the other collected measurements.
  Stable absent (i.e., all measurements 'No), Stable present (i.e., all measurements 'Yes'), Improved (i.e., last measurement collected as 'No' and baseline 'Yes'), Worsened (i.e., last measurement collected 'Yes' and baseline 'No').
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  Stable absent; q12w fluid free - No | 39
  Stable present; q12w fluid free - No | 32
  Improved; q12w fluid free - No | 20
  Worsened; q12w fluid free - No | 2

5. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Sub-retinal Pigment Epithelium (Sub-RPE) Fluid - Patients Classified as q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  Stable absent; q12w fluid free - Yes | 12
  Stable present; q12w fluid free - Yes | 7
  Improved; q12w fluid free - Yes | 8
  Worsened; q12w fluid free - Yes | 0

6. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Subretinal Hyperreflective Material (SHRM) - Patients Classified as Not q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  Stable absent; q12w fluid free - No | 41
  Stable present; q12w fluid free - No | 33
  Improved; q12w fluid free - No | 7
  Worsened; q12w fluid free - No | 12

7. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Subretinal Hyperreflective Material (SHRM) - Patients Classified as q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  Stable absent; q12w fluid free - Yes | 11
  Stable present; q12w fluid free - Yes | 7
  Improved; q12w fluid free - Yes | 4
  Worsened; q12w fluid free - Yes | 5

8. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Outer Retinal Tubulation (ORT) - Patients Classified as Not q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  Stable absent; q12w fluid free - No | 84
  Stable present; q12w fluid free - No | 1
  Improved; q12w fluid free - No | 3
  Worsened; q12w fluid free - No | 5

9. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Outer Retinal Tubulation (ORT) - Patients Classified as q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  Stable absent; q12w fluid free - Yes | 25
  Stable present; q12w fluid free - Yes | 2
  Improved; q12w fluid free - Yes | 0
  Worsened; q12w fluid free - Yes | 0

10. Primary Outcome: Potential Predictor Factors of Fluid-free Response: External Limiting Membrane (ELM) Integrity Loss in Center 1 mm - Patients Classified as Not q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  Stable absent; q12w fluid free - No | 25
  Stable present; q12w fluid free- No | 43
  Improved; q12w fluid free - No | 11
  Worsened; q12w fluid free - No | 14

11. Primary Outcome: Potential Predictor Factors of Fluid-free Response: External Limiting Membrane (ELM) Integrity Loss in Center 1 mm - Patients Classified as q12w Fluid-free
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  Stable absent; q12w fluid free - Yes | 8
  Stable present; q12w fluid free - Yes | 13
  Improved; q12w fluid free - Yes | 3
  Worsened; q12w fluid free - Yes | 3

12. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Type of Pigment Epithelium Detachment (PED) - Patients Classified as Not q12w Fluid-free
Description: As assessed by Spectral Domain Optical Coherence Tomography (SD-OCT).
  Percentages were computed on Safety Population within 'No' and 'Yes' groups according to q12w fluid free.
  * Stable Fibrovascular only (i.e., all measurements 'Fibrovascular only').
  * Stable not only fibrovascular (i.e., all measurements 'Predominantly fibrovascular' or 'Predominantly serous' or 'Drusenoid Pigment Epithelial Detachment (PED)').
  * From not only fibrovascular to Fibrovascular only (i.e., last measurement collected 'Fibrovascular only' and baseline 'Predominantly fibrovascular' or 'Predominantly serous' or 'Drusenoid PED').
  * From Fibrovascular only to not only fibrovascular (i.e., last measurement collected 'Predominantly fibrovascular' or 'Predominantly serous' or 'Drusenoid PED' and baseline 'Fibrovascular only').
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 93
Participants
  Stable Fibrovascular only; q12w fluid free - No | 38
  Stable not only fibrovascular; q12w fluid free - No | 28
  From not only fibrovascular to Fibrovascular only; q12w fluid free - No | 24
  From Fibrovascular only to not only fibrovascular; q12w fluid free - No | 3

13. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Type of Pigment Epithelium Detachment (PED) - Patients Classified as q12w Fluid-free
Description: as for outcome 12
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Participants
  Stable Fibrovascular only; q12w fluid free - Yes | 13
  Stable not only fibrovascular; q12w fluid free - Yes | 7
  From not only fibrovascular to Fibrovascular only; q12w fluid free - Yes | 7
  From Fibrovascular only to not only fibrovascular; q12w fluid free - Yes | 0

14. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Percentage Changes in Central Subfield Thickness (CST) From Baseline at Week 16 - Patients Classified as q12w Fluid-free
Description: As assessed by Spectral Domain Optical Coherence Tomography (SD-OCT).
  Mean (SD) was computed on the Safety Population within 'No' and 'Yes' groups according to q12w fluid free.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
Percentage change | -36.4 (16.85)

15. Primary Outcome: Potential Predictor Factors of Fluid-free Response: Percentage Changes in Central Subfield Thickness (CST) From Baseline at Week 16 - Patients Classified as Not q12w Fluid-free
Description: as for outcome 14
Time Frame: Baseline, Week 16
Population: Full Analysis Set - includes all patients who received at least one dose of the study drug and who were classified as not q12w fluid-free and with a valid measurement without a protocol deviation with impact. (N=92). (Excludes patients with protocol deviations.)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 92
Percentage change | -31.7 (18.28)

16. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Branching Vessels
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD)
  The morphology of the Neovascularization (CNV) complex was evaluated qualitatively by assessing the presence/absence of branching vessels. The presence of tiny vessels branching from bigger vessels is indicative of an active CNV lesion.
  UNG/P = Ungradable due to pathology UNG/Q = Ungradable due to Quality
Time Frame: Baseline, Week 16, Week 48
Population: Full Analysis Set - includes all patients who received at least one dose of the study drug with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  Branching Vessels - Increased from prior - Week 16 | 11
  Branching Vessels - Increased from prior - Week 48 (n=91): number analyzed (Participants) | 91
  Branching Vessels - Increased from prior - Week 48 (n=91) | 4
  Branching Vessels - Decreased from prior - Week 16 | 2
  Branching Vessels - Decreased from prior - Week 48 (n=91): number analyzed (Participants) | 91
  Branching Vessels - Decreased from prior - Week 48 (n=91) | 11
  Branching Vessels - Stable - Week 16 | 26
  Branching Vessels - Stable - Week 48 (n=91): number analyzed (Participants) | 91
  Branching Vessels - Stable - Week 48 (n=91) | 20
  Branching Vessels - UNG/P - Week 16 | 9
  Branching Vessels - UNG/P - Week 48 (n=91): number analyzed (Participants) | 91
  Branching Vessels - UNG/P - Week 48 (n=91) | 21
  Branching Vessels - UNG/Q - Week 16 | 66
  Branching Vessels - UNG/Q - Week 48 (n=91): number analyzed (Participants) | 91
  Branching Vessels - UNG/Q - Week 48 (n=91) | 35

17. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Change From Baseline of Total CNV Lesion Area (mm*2)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD).
  The total Basal Choroidal Neovascularization (CNV) lesion area (mm^2) and greatest linear diameter of lesion (mm) are the parameters related to CNV flow size.
Time Frame: Baseline, Week 16, Week 48
Population: Full Analysis Set - includes all patients with a CNV lesion who received at least one dose of the study drug with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
mm^2
  Week 16 (n=27) | 0.476 (1.0012)
  Week 48 (n=20): number analyzed (Participants) | 20
  Week 48 (n=20) | 0.533 (0.9053)

18. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Change From Baseline of Choroidal Neovascularization (CNV) Vascular Density (%)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD).
  The Choroidal Neovascularization (CNV) vascular density (%) is calculated as a ratio of the area occupied by vessels and the total area of the lesion and multiplied by 100.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: % CNV Vascular Density
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 9
% CNV Vascular Density
  Week 16 | 1.326 (35.6003)
  Week 48 (n=8): number analyzed (Participants) | 8
  Week 48 (n=8) | 29.900 (52.3079)

19. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Change From Baseline of Lesion Greatest Linear Diameter (mm)
Description: as for outcome 17
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 27
mm
  Week 16 | -0.211 (0.5416)
  Week 48 (n=20): number analyzed (Participants) | 20
  Week 48 (n=20) | -0.147 (0.5837)

20. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Peripheral Anastomotic Arcades
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD).
  The morphology of the Choroidal Neovascularization (CNV) complex was evaluated qualitatively by assessing the peripheral anastomotic arcades. The presence of peripheral anastomotic arcades at the vessel termini is indicative of an active CNV lesion.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 25
Participants
  No at Baseline and No at Week 16 | 14
  Yes at Baseline and No at Week 16 | 1
  No at Baseline and Yes at Week 16 | 4
  Yes at Baseline and Yes at Week 16 | 6
  No at Baseline and No at Week 48 (n=21): number analyzed (Participants) | 21
  No at Baseline and No at Week 48 (n=21) | 7
  Yes at Baseline and No at Week 48 (n=21): number analyzed (Participants) | 21
  Yes at Baseline and No at Week 48 (n=21) | 2
  No at Baseline and Yes at Week 48 (n=21): number analyzed (Participants) | 21
  No at Baseline and Yes at Week 48 (n=21) | 8
  Yes at Baseline and Yes at Week 48 (n=21): number analyzed (Participants) | 21
  Yes at Baseline and Yes at Week 48 (n=21) | 4

21. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Vascular Loops
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD).
  The morphology of the Choroidal Neovascularization (CNV) complex was evaluated qualitatively by assessing the vascular loops. The presence of vascular loops is indicative of an active CNV lesion.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 26
Participants
  No at Baseline and No at Week 16 | 12
  Yes at Baseline and No at Week 16 | 1
  No at Baseline and Yes at Week 16 | 3
  Yes at Baseline and Yes at Week 16 | 10
  No at Baseline and No at Week 48 (n=22): number analyzed (Participants) | 22
  No at Baseline and No at Week 48 (n=22) | 4
  Yes at Baseline and No at Week 48 (n=22): number analyzed (Participants) | 22
  Yes at Baseline and No at Week 48 (n=22) | 3
  No at Baseline and Yes at Week 48 (n=22): number analyzed (Participants) | 22
  No at Baseline and Yes at Week 48 (n=22) | 7
  Yes at Baseline and Yes at Week 48 (n=22): number analyzed (Participants) | 22
  Yes at Baseline and Yes at Week 48 (n=22) | 8

22. Secondary Outcome: Change in Optical Coherence Tomography (OCTA) Features Baseline up to Week 48 - Dark Halo
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD).
  The morphology of the Choroidal Neovascularization (CNV) complex was evaluated qualitatively by assessing the dark halo. The presence of dark halo is considered a region of choriocapillaris alteration corresponding to local flow impairment and is indicative of an active CNV lesion.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 17
Participants
  No at Baseline and No at Week 16 (n=15): number analyzed (Participants) | 15
  No at Baseline and No at Week 16 (n=15) | 9
  Yes at Baseline and No at Week 16 (n=15): number analyzed (Participants) | 15
  Yes at Baseline and No at Week 16 (n=15) | 2
  No at Baseline and Yes at Week 16 (n=15): number analyzed (Participants) | 15
  No at Baseline and Yes at Week 16 (n=15) | 0
  Yes at Baseline and Yes at Week 16 (n=15): number analyzed (Participants) | 15
  Yes at Baseline and Yes at Week 16 (n=15) | 4
  No at Baseline and No at Week 48 (n=17) | 6
  Yes at Baseline and No at Week 48 (n=17) | 5
  No at Baseline and Yes at Week 48 (n=17) | 2
  Yes at Baseline and Yes at Week 48 (n=17) | 4

23. Secondary Outcome: Spectral Domain Optical Coherence Tomography (SD-OCT) Features Baseline up to Week 48 - Pigment Epithelial Detachment (PED)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD)
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 120
Participants
  Yes - Baseline | 120
  Yes - Week 16 (n=114): number analyzed (Participants) | 114
  Yes - Week 16 (n=114) | 114
  Yes - Week 48 (n=93): number analyzed (Participants) | 93
  Yes - Week 48 (n=93) | 92
  Missing - Week 48 (n=93): number analyzed (Participants) | 93
  Missing - Week 48 (n=93) | 1

24. Secondary Outcome: Spectral Domain Optical Coherence Tomography (SD-OCT) Features Baseline up to Week 48 - Central Subfield Thickness (CST) (μm)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  The central retina thickness (CRT) evaluated in this study represents the average retinal thickness of the circular area within 1 mm diameter around the foveal center and was called Center Subfield Thickness (CST), also known as foveal thickness.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 120
micrometers
  Baseline | 482.6 (177.40)
  Week 16 (n=114): number analyzed (Participants) | 114
  Week 16 (n=114) | 309.2 (107.69)
  Week 48 (n=93): number analyzed (Participants) | 93
  Week 48 (n=93) | 307.9 (118.05)

25. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative OCTA parameters of wet Age-related Macular Degeneration (wAMD)
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 76
micrometers
  Week 16 | -188.4 (142.79)
  Week 48 (n=60): number analyzed (Participants) | 60
  Week 48 (n=60) | -197.6 (152.63)

26. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - Intraretinal Fluid (IRF) Cystoid Edema
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  IRF is the fluid that accumulates within the neurosensory retina due to the disruption of the external limiting membrane (ELM)-photoreceptor complex in the outer retina by the active Choroidal Neovascularization (CNV) membrane.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  No at Baseline and No at Week 16 | 46
  Yes at Baseline and No at Week 16 | 38
  No at Baseline and Yes at Week 16 | 4
  Yes at Baseline and Yes at Week 16 | 26
  No at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and No at Week 48 (n=92) | 40
  Yes at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and No at Week 48 (n=92) | 30
  No at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and Yes at Week 48 (n=92) | 1
  Yes at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and Yes at Week 48 (n=92) | 21

27. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - Subretinal Fluid (SRF)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  SRF is the fluid that commonly accumulates between the neurosensory retina and the retinal pigment epithelium (RPE) due to the profuse leakage from blood vessels of the Choroidal Neovascularization (CNV) complex.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  No at Baseline and No at Week 16 | 7
  Yes at Baseline and No at Week 16 | 75
  No at Baseline and Yes at Week 16 | 1
  Yes at Baseline and Yes at Week 16 | 31
  No at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and No at Week 48 (n=92) | 6
  Yes at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and No at Week 48 (n=92) | 57
  No at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and Yes at Week 48 (n=92) | 0
  Yes at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and Yes at Week 48 (n=92) | 29

28. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - Sub Retinal Pigment Epithelium (Sub RPE) Fluid
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  Sub-RPE fluid, i.e., the fluid that accumulates under the RPE, thus often leading to Pigment Epithelial Detachments (PEDs).
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  No at Baseline and No at Week 16 | 49
  Yes at Baseline and No at Week 16 | 26
  No at Baseline and Yes at Week 16 | 1
  Yes at Baseline and Yes at Week 16 | 38
  No at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and No at Week 48 (n=92) | 36
  Yes at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and No at Week 48 (n=92) | 26
  No at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and Yes at Week 48 (n=92) | 2
  Yes at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and Yes at Week 48 (n=92) | 28

29. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - Subretinal Hyperreflective Material (SHRM)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  SHRM, i.e., a poorly defined, medium-to-hyperreflective mass between the neurosensory layers and the sub retinal pigment epithelium (RPE) on SD-OCT, which is indicative of the neurovascular membrane, particularly in type II Choroidal Neovascularization (CNV) lesions, and of disciform scar formation
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  No at Baseline and No at Week 16 | 50
  Yes at Baseline and No at Week 16 | 11
  No at Baseline and Yes at Week 16 | 16
  Yes at Baseline and Yes at Week 16 | 37
  No at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and No at Week 48 (n=92) | 45
  Yes at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and No at Week 48 (n=92) | 14
  No at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and Yes at Week 48 (n=92) | 8
  Yes at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and Yes at Week 48 (n=92) | 25

30. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - Outer Retinal Tubulation (ORT)
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  ORT, i.e., branching tubular structures located in the outer nuclear layer of the retina, which seems to be indicative of a rearrangement of degenerating photoreceptors in a variety of retinal diseases, including wAMD. On SD-OCT, ORT appears as well-defined round or ovoid hyporeflective spaces with hyperreflective borders.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 114
Participants
  No at Baseline and No at Week 16 | 103
  Yes at Baseline and No at Week 16 | 3
  No at Baseline and Yes at Week 16 | 5
  Yes at Baseline and Yes at Week 16 | 3
  No at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and No at Week 48 (n=92) | 77
  Yes at Baseline and No at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and No at Week 48 (n=92) | 3
  No at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  No at Baseline and Yes at Week 48 (n=92) | 10
  Yes at Baseline and Yes at Week 48 (n=92): number analyzed (Participants) | 92
  Yes at Baseline and Yes at Week 48 (n=92) | 2

31. Secondary Outcome: Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Features From Baseline up to Week 48 - External Limiting Membrane (ELM) Integrity Loss
Description: Evaluate the effect of brolucizumab on the evolution of qualitative and quantitative SCD-OCT parameters of wet Age-related Macular Degeneration (wAMD).
  Status of the ELM as an indicator of retinal integrity was evaluated focusing on ELM integrity loss in center 1 mm (i.e., considering the central 1 x 1-mm subfield).
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 113
Participants
  No at Baseline and No at Week 16 | 30
  Yes at Baseline and No at Week 16 | 14
  No at Baseline and Yes at Week 16 | 15
  Yes at Baseline and Yes at Week 16 | 54
  No at Baseline and No at Week 48 (n=91): number analyzed (Participants) | 91
  No at Baseline and No at Week 48 (n=91) | 24
  Yes at Baseline and No at Week 48 (n=91): number analyzed (Participants) | 91
  Yes at Baseline and No at Week 48 (n=91) | 9
  No at Baseline and Yes at Week 48 (n=91): number analyzed (Participants) | 91
  No at Baseline and Yes at Week 48 (n=91) | 15
  Yes at Baseline and Yes at Week 48 (n=91): number analyzed (Participants) | 91
  Yes at Baseline and Yes at Week 48 (n=91) | 43

32. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) From Baseline up to Week 48
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of >= 34 ETDRS letters (Snellen equivalent 20/200) at Screening / Baseline in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
  Last observation carried forward (LOCF) was used for the imputation of missing values.
Time Frame: Baseline, Week 16, Week 48
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: Letters read
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 120
Letters read
  Week 16 | 4.0 [0.0 to 10.0]
  Week 48 | 5.5 [-0.5 to 12.0]

33. Secondary Outcome: Number of Patients With Fluid Resolution of the Study Eye
Description: Evaluate the effect of brolucizumab on sustained dryness from Baseline to Week 48.
  Among patients with fluid present at Baseline, patients with fluid resolution were identified in case of absence of IRF and SRF and patients without fluid resolution were categorized in 'only IRF present', 'only SRF present', 'both IRF and SRF present' at each post-baseline timepoint.
  IRF = Intraretinal Fluid SRF = Subretinal Fluid
Time Frame: Week 16, Week 48
Population: Full Analysis Set - includes all patients with fluid present at Baseline who received at least one dose of the study drug with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 113
Participants
  Patients with fluid resolution - Week 16 | 64
  Patients without fluid resolution - Week 16 | 49
  Patients without fluid resolution - Only IRF present - Week 16 (n=49): number analyzed (Participants) | 49
  Patients without fluid resolution - Only IRF present - Week 16 (n=49) | 18
  Patients without fluid resolution - Only SRF present - Week 16 (n=49): number analyzed (Participants) | 49
  Patients without fluid resolution - Only SRF present - Week 16 (n=49) | 19
  Patients without fluid resolution - Both IRF and SRF present - Week 16 (n=49): number analyzed (Participants) | 49
  Patients without fluid resolution - Both IRF and SRF present - Week 16 (n=49) | 12
  Patients with fluid resolution - Week 48 (n=92): number analyzed (Participants) | 92
  Patients with fluid resolution - Week 48 (n=92) | 49
  Unknown- Week 48 (n=92): number analyzed (Participants) | 92
  Unknown- Week 48 (n=92) | 1
  Patients without fluid resolution - Week 48 (n=92): number analyzed (Participants) | 92
  Patients without fluid resolution - Week 48 (n=92) | 42
  Patients without fluid resolution - Only IRF present - Week 48 (n=42): number analyzed (Participants) | 42
  Patients without fluid resolution - Only IRF present - Week 48 (n=42) | 13
  Patients without fluid resolution - Only SRF present - Week 48 (n=42): number analyzed (Participants) | 42
  Patients without fluid resolution - Only SRF present - Week 48 (n=42) | 20
  Patients without fluid resolution - Both IRF and SRF present - Week 48 (n=42): number analyzed (Participants) | 42
  Patients without fluid resolution - Both IRF and SRF present - Week 48 (n=42) | 9

34. Secondary Outcome: Sustained Dryness of the Study Eye - Kaplan-Meier Estimates - Median Time to the Achievement of Sustained Dryness
Description: Evaluate the effect of brolucizumab on sustained dryness from Baseline to Week 48.
  Patients who achieved sustained dryness were identified considering those with fluid resolution for at least 2/3 consecutive visits.
  Median time to the achievement of sustained dryness was calculated by the Kaplan-Meier method.
  Sustained dryness of the study eye, is defined by the absence of IRF and SRF for at least 2 consecutive visits and for at least 3 consecutive visits.
  IRF = Intraretinal Fluid SRF = Subretinal Fluid
Time Frame: Up to Week 48
Population: Full Analysis Set - includes all patients with fluid present at baseline and who received at least one dose of the study drug with a valid measurement without a protocol deviation with impact.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 119
weeks | 16.43 [12.86 to 31.00]

35. Secondary Outcome: Cumulative Incidence of Patients With Sustained Dryness of the Study Eye
Description: Evaluate the effect of brolucizumab on sustained dryness from Baseline to Week 48.
  Sustained dryness of the study eye, is defined by the absence of IRF and SRF for at least 2 consecutive visits and for at least 3 consecutive visits.
  IRF = Intraretinal Fluid SRF = Subretinal Fluid
Time Frame: Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 119
Participants
  Patients with sustained dryness - Week 8 | 36
  Patients with sustained dryness - Week 12 | 54
  Patients with sustained dryness - Week 16 | 64
  Patients with sustained dryness - Week 20 | 68
  Patients with sustained dryness - Week 24 | 68
  Patients with sustained dryness - Week 28 | 68
  Patients with sustained dryness - Week 32 | 73
  Patients with sustained dryness - Week 36 | 76
  Patients with sustained dryness - Week 40 | 77
  Patients with sustained dryness - Week 44 | 77
  Patients with sustained dryness - Week 48 | 78

36. Secondary Outcome: Determinants in the Investigator's Choice of Brolucizumab Dosing Regimen (q8w) at Week 16
Description: Evaluate the reasons underlying the Investigators' choice of brolucizumab treatment regimen (q8w)
  BVCA=Best-Corrected Visual Acuity, CFP=Color Fundus Photography; CNV=Choroidal Neovascularization; FA=Fluorescein Angiography; ICGA=IndoCyanine Green Angiography; OCTA=Optical Coherence Tomography Angiography; SD-OCT=Spectral Domain Optical Coherence Tomography
Time Frame: Up to Week 16
Population: Full Analysis Set - iincludes Patients who performed Week 16 and still on treatment of brolucizumab dosing regimen (q8w) with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 42
Participants
  Intraretinal fluid (IRF) at SD-OCT | 17
  Subretinal fluid (SRF) at SD-OCT | 21
  Central Subfield Thickness (CST) at SD-OCT | 15
  Best-corrected visual acuity (BCVA) | 13
  Subretinal pigment epithelium (sub-RPE) fluid at SD-OCT | 4
  Central Retinal Thickness (CRT) | 4
  Subretinal hyperreflective material (SHRM) at Domain Optical Coherence Tomography. (SD-OCT) | 6
  Retina Pigment Epithelial Detachment volume at SD-OCT | 3
  CNV size at OCTA | 2
  Hemorrhage at CFP | 2
  Vessel morphology at OCTA | 2
  Vessel density at OCTA | 3
  Other - investigator's discretion | 2
  Leakage at FA/ICGA | 0

37. Secondary Outcome: Determinants in the Investigator's Choice of Brolucizumab Dosing Regimen (q12w) at Week 16
Description: Evaluate the reasons underlying the Investigators' choice of brolucizumab treatment regimen (q12w)
  BVCA=Best-Corrected Visual Acuity, CFP=Color Fundus Photography; CNV=Choroidal Neovascularization; FA=Fluorescein Angiography; ICGA=IndoCyanine Green Angiography; OCTA=Optical Coherence Tomography Angiography; SD-OCT=Spectral Domain Optical Coherence Tomography
Time Frame: Up to Week 16
Population: Full Analysis Set - includes Patients who performed Week 16 and still on treatment of brolucizumab dosing regimen (q12w) with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 68
Participants
  Intraretinal fluid (IRF) at SD-OCT | 46
  Subretinal fluid (SRF) at SD-OCT | 41
  Central Subfield Thickness (CST) at SD-OCT | 35
  BCVA | 29
  Subretinal pigment epithelium (sub-RPE) fluid at SD-OCT | 26
  Central Retinal Thickness (CRT) | 26
  Subretinal hyperreflective material (SHRM) at SD-OCT | 22
  Retina Pigment Epithelial Detachment volume at SD-OCT | 19
  CNV size at OCTA | 18
  Hemorrhage at CFP | 17
  Vessel morphology at OCTA | 13
  Vessel density at OCTA | 11
  Other - investigator's discretion | 11
  Leakage at FA/ICGA | 0

38. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Scores
Description: Evaluate anxiety/depression in patients with wAMD treated with brolucizumab. The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale that generates ordinal data. Seven items relate to anxiety and seven relate to depression. This patient-reported outcome measure was specifically developed to avoid reliance on anxiety/depression aspects which are also common somatic symptoms of illness, such as fatigue and insomnia or hypersomnia. Calculations of scores: each item is rated on a 4-point scale. The HADS consists of two sub-scores: the HAD-A for anxiety and HAD-D for depression. Each sub-score ranges from 0 to 21 points: scores ≥11 indicate the presence of an anxious or depressive disorder, scores between 8-10 points are borderline abnormal, and scores ≤7 indicate that an anxious or depressive disorder is not present.
Time Frame: Up to Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 96
Scores on a scale
  HAD-A - Absolute change from baseline at Week 48 | -0.78 (3.258)
  HAD-D - Absolute change from baseline at Week 48 | -0.10 (3.049)

39. Secondary Outcome: Change in European Quality of Life-5D-5L (EQ-5D-5L) Scores
Description: Evaluate quality of life in patients with wAMD treated with brolucizumab. The EQ-5D-5L is a standardized widely used instrument for measuring generic health status. It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels. i.e. no problems, slight problems, moderate problems, severe problems and extreme problems, corresponding to digit numbers ranging from 1 to 5. The EQ-5D-5L total score is determined through a Visual Analogue Scale (VAS) and ranges from 0 to 100 with higher scores indicative of a better health status.
Time Frame: Baseline, Week 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 96
Scores on a scale | 0.00 (0.147)

40. Secondary Outcome: Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject
Time Frame: AEs are reported from first dose of study treatment until 4 weeks after last treatment, for a maximum time frame of approx. 48 weeks.
Population: Safety Set - includes all patients who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 122
Participants
  Patients with TEAEs | 59
  Patients with Serious TEAEs | 14
  Patients with Ocular TEAEs | 33
  Patients with non-ocular TEAEs | 40
  Patients with suspected drug-related TEAEs | 13
  Patients with TEAEs related to Ocular injection procedure | 4
  Patients with TEAEs leading to temporary interruption of treatment | 2
  Patients with TEAEs leading to withdrawn of treatment | 15
  Patients with TEAEs leading to study discontinuation | 7
  Patients with TEAEs with fatal outcome | 0

41. Secondary Outcome: Ocular Treatment Emergent Adverse Events - Study Eye
Description: as for outcome 40
Time Frame: as for outcome 40
Population: Safety Set - includes all patients who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 122
Participants
  Patients with Ocular TEAEs | 25
  Patients with Serious Ocular TEAEs | 1
  Patients with suspected drug-related Ocular TEAEs | 11
  Patients with Ocular TEAEs related to Ocular injection procedure | 3
  Patients with Ocular TEAEs leading to temporary interruption of treatment | 1
  Patients with Ocular TEAEs leading to withdrawn of treatment | 10
  Patients with Ocular TEAEs leading to study discontinuation | 5
  Patients with Ocular TEAEs with fatal outcome | 0

42. Secondary Outcome: Ocular Treatment Emergent Adverse Events - by System Organ Class (SOC) and Preferred Term (PT)
Description: as for outcome 40
Time Frame: as for outcome 40
Population: Safety Set - includes all patients who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 122
Participants
  Eye disorders | 30
  -Cataract | 3
  -Conjunctival haemorrhage | 1
  -Eye haemorrhage | 1
  -Eye inflammation | 2
  -Iridocyclitis | 1
  -Macular degeneration | 1
  -Macular detachment | 1
  -Macular fibrosis | 2
  -Macular hole | 3
  -Maculopathy | 1
  -Neovascular age-related macular degeneration | 3
  -Ocular hypertension | 2
  -Retinal haemorrhage | 1
  -Retinal occlusive vasculitis | 1
  -Retinal pigment epithelial tear | 3
  -Retinal tear | 2
  -Retinal vascular disorder | 1
  -Retinal vasculitis | 1
  -Uveitis | 1
  -Vision blurred | 1
  -Visual impairment | 1
  -Vitreous floaters | 1
  -Vitritis | 5

ADVERSE EVENTS:
Time Frame: Adverse Events are reported from first dose of study treatment until 4 weeks after last treatment, for a maximum time frame of approx. 48 weeks.
Arm/Group | Brolucizumab 6 mg
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 14/122
Other Adverse Events (participants affected / at risk) | 52/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6 mg (N=122)
Acute myocardial infarction (Cardiac disorders) | 1
Retinal occlusive vasculitis- Study eye (Eye disorders) | 1
Uveitis- Study eye (Eye disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Condition aggravated (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Acute undifferentiated leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6 mg (N=122)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Defect conduction intraventricular (Cardiac disorders) | 1
Diastolic dysfunction (Cardiac disorders) | 1
Cataract- Both (Eye disorders) | 1
Cataract- Fellow eye (Eye disorders) | 1
Cataract- Study eye (Eye disorders) | 2
Conjunctival haemorrhage- Study eye (Eye disorders) | 1
Eye haemorrhage- Fellow eye (Eye disorders) | 1
Eye inflammation- Study eye (Eye disorders) | 2
Iridocyclitis- Study eye (Eye disorders) | 1
Macular degeneration- Fellow eye (Eye disorders) | 1
Macular detachment- Fellow eye (Eye disorders) | 1
Macular fibrosis- Study eye (Eye disorders) | 2
Macular hole- Study eye (Eye disorders) | 3
Maculopathy- Study eye (Eye disorders) | 1
Neovascular age-related macular degeneration- Fellow eye (Eye disorders) | 3
Ocular hypertension- Both (Eye disorders) | 1
Ocular hypertension- Study eye (Eye disorders) | 1
Retinal haemorrhage- Study eye (Eye disorders) | 1
Retinal pigment epithelial tear- Study eye (Eye disorders) | 3
Retinal tear- Study eye (Eye disorders) | 2
Retinal vascular disorder- Study eye (Eye disorders) | 1
Retinal vasculitis- Study eye (Eye disorders) | 1
Vision blurred- Study eye (Eye disorders) | 1
Visual impairment- Study eye (Eye disorders) | 1
Vitreous floaters- Study eye (Eye disorders) | 1
Vitritis- Study eye (Eye disorders) | 5
Aphthous ulcer (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 13
Conjunctivitis bacterial- Both (Infections and infestations) | 1
Conjunctivitis- Study eye (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Blood pressure abnormal (Investigations) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arachnoid cyst (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Gliosis (Nervous system disorders) | 1
Nystagmus- Fellow eye (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis- Fellow eye (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Vasculitis- Study eye (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT04774926/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04774926/SAP_001.pdf